CLINICAL TRIAL: NCT01330862
Title: Epidemiological Study to Describe NSCLC Clinical Management Patterns in MENA. Lung-EPICLIN/ KSA
Brief Title: Epidemiological Study to Describe Non-small-cell Lung Carcinoma (NSCLC) Clinical Management Patterns in MENA. Lung-EPICLIN/ KSA
Acronym: EPICLIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-MENA-SA-IRS-2010/01
Record Dates: First submitted 2011-03-30; First posted 2011-04-07 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: NSCLC Patient Characteristics
Keywords: patient outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is to provide accurate, reliable information on NSCLC clinical management across MENA (Middle East North Africa) countries in order to detect unmet medical needs of this disease, it is a purely observational study; therefore patients are not assigned to a particular therapeutic strategy beforehand by a protocol. Treatment will be according to current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NSCLC diagnosis (e.g. bronchoscope or FNAB), all stages, men and women, attending the responsible department of treating this type of patients for the first time between April 1st 2011 and March 31 2012, for PRO sub-sample: ability to read and write since they will be asked to participate in the PRO part of the study. Selection will not be based on the disease stage of each patient, in order to avoid a selection bias

Exclusion Criteria:

* According to the study design there will not be any exclusion criteria in order to provide a high validity and to obtain the most accurate real daily practice information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All NSCLC patients attending the responsible department of treating this type of patients (e.g. Oncology Department) for the first time (regardless of whether the patient is diagnosed with locally, advanced or metastatic disease) at the participating sites from the first of April 2011 to the end of September 2011
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Abdul Rahman Jazieh, Study Chair — King Fahad National Guard Hospital; Dr. Ahmed Abdulwarith, Principal Investigator — King Fahad Specialist Hospital; Dr. Rasha Moastafa, Principal Investigator — King Fahad Medical City; Dr. Sherif Wafa, Principal Investigator — Prince Faisal Bin Bander oncology centre; Dr. Maged Mansour, Principal Investigator — Dr. Erfan & Bagedo Hospital; Dr. Mohamed Rahhal, Principal Investigator — King Fahad Specialist Hospital
Locations (4):
- Saudi Arabia (4):
  - Research Site, Qassim, Central
  - Research Site, Riyadh, Central
  - Research Site, Dammam, Eastern Province
  - Research Site, Jeddah, Western